CLINICAL TRIAL: NCT01812018
Title: An Open-label, Single-arm, Phase II Study to Assess the Efficacy and Safety of Endostar® (Recombinant Human Endostatin Injection) Plus Gemcitabine and Docetaxel in Treatment of Soft Tissue Sarcoma Patients With Pulmonary Metastases
Brief Title: Endostar + GT in Pulmonary Metastases of Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peng Yuan (Unknown)
Responsible Party: Sponsor-Investigator, Peng Yuan, Associate Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-SAR-001
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; Pulmonary metastases
MeSH Terms: conditions — Sarcoma | interventions — endostar protein; Endostatins; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar (Experimental): Endostar, Gemcitabine, Docetaxel
  Interventions: Drug: Endostar; Drug: Gemcitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Endostar — Endostar administered at 7.5 mg/m2, intravenously (IV), on Day 1-14 every 21 days for up to 4-6 consecutive cycles
  Other Names: Recombinant Human Endostatin Injection
Drug: Gemcitabine — Gemcitabine administered at 1000 mg/m2, intravenously (IV), on Day 1 and Day 8, every 21 days for up to 4-6 consecutive cycles
Drug: Docetaxel — Docetaxel administered at 75 mg/m2, intravenously (IV), on Day 2, every 21 days for up to 4-6 consecutive cycles

SUMMARY:
The purpose of this exploratory phase II study is to assess the effectiveness and safety profile of Endostar®(Recombinant Human Endostatin Injection) plus Gemcitabine and Docetaxel in treatment of soft tissue sarcoma patients with pulmonary metastases.

DETAILED DESCRIPTION:
Anticipated 30 subjects will be enrolled to receive Endostar, Gemcitabine and Docetaxel. Endostar at a dosage of 7.5 mg/m2 will be administered on Day 1-14 of each cycle. Gemcitabine (1000 mg/m2) will be administered on Day 1 and Day 8 of each cycle. Docetaxel (75 mg/m2) will be administered on Day 2 of each cycle. An individual cycle of therapy will be defined as a 3-week (21-day) period. Cycles will be repeated every 3 weeks. Multiple cycles may be administered until the subject is PD or until a maximum of 6 cycles. Time-to-progression (TTP) will be assessed using the Kaplan Meier method. Overall response rate (ORR) as well as individual categories of response (CR, PR, SD, and PD) will be determined using RECIST (v1.1). Evaluation of 1- and 2-year overall survival will also be performed. Safety measures will be recorded using the NCI-CTCAE (v4.0).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years, male or female.
* ECOG performance status <=2.
* Life expectancy >= 3 months.
* Histologically or cytologically confirmed soft tissue sarcoma (GIST excluded).
* Patients must have had a prior anthracycline and/or ifosfamide in either the adjuvant or metastatic setting but not more than one regimen.
* At least one measurable pulmonary metastasis tumor lesions according to RECIST 1.1 criteria.
* Laboratory values: Hemoglobin (Hb) >= 90 g/L and no blood transfusion within 14 days, Absolute neutrophil count (ANC) >= 1.5 x 10^9/L, Platelet (Plt)>= 80 x 10^9/L, Total Bilirubin (Tbil)=< 1.5 x upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN or =< 5 x ULN if liver metastases are present, Serum creatinine (Cr) =< 1.0 x ULN, Endogenous creatinine clearance (Ccr)> 50 mL/min (Cockcroft-Gault).
* Women of child bearing potential must have a negative serum or urine pregnancy test within 7 days before enrollment and be willing to use effective contraception during study and for 8 weeks after last IMP administration.
* Willingness to participate in study and sign informed consent form.

Exclusion Criteria:

* Females who are pregnant or breastfeeding or have Childbearing potential unwilling to use effective contraception.
* Prior therapy with Gemcitabine, Docetaxel and Endostar.
* Subjects participating in other clinical trials within 4 weeks before enrollment.
* Accompanied by rapid progress of organ invasions, e.g.lesion areas are great than one half of liver or lung or have liver dysfunction.
* Uncontrolled central nervous system disorder or psychiatric illness.
* Current, serious, clinically significant cardiac arrhythmias, symptomatic congestive heart failure, myocardial infarction before enrollment.
* Patients with abnormal bone marrow function: ANC < 1.5 x 10^9/L, Plt < 75 x 10^9/L, Hb < 90g/L.
* Patients with renal dysfunction: Cr > 1.5 x ULN.
* Patients with liver dysfunction: Tbil > 1.5 x ULN.
* Uncontrolled brain metastases.
* Unwillingness or inability to comply with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Time-to-Progression | Approximately 2 years
  Time to progression is defined as time from first study treatment dose to the progression disease.

SECONDARY OUTCOMES:
Overall Response Rate | Approximately 2 years
Evaluate 1-year and 2-year overall survival rates | Approximately 2 years
Safety measures | Approximately 3 years
  Adverse events, Clinical and laboratory data including physical examinations, vital signs, ECG results, Use of concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China